CLINICAL TRIAL: NCT03425292
Title: A Longitudinal Assessment of Tumor Evolution in Patients With Brain Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Principal Investigator, Santosh Kesari, Professor, Neurosciences, Saint John's Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JWCI-17-0801
Record Dates: First submitted 2018-01-21; First posted 2018-02-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Newly Diagnosed High Grade Glioma
Keywords: immunotherapy; nivolumab; ipilimumab; bevcizumab; temozolomide
MeSH Terms: interventions — Temozolomide; Nivolumab; Ipilimumab; Bevacizumab; Lomustine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1 SOC (closed to enrollment) (Active Comparator): Standard conformal brain radiation therapy with concurrent and adjuvant temozolomide
  Interventions: Drug: Temozolomide; Radiation: conformal brain radiation therapy
- 2 Nivo (Experimental): Nivolumab
  Interventions: Drug: Nivolumab monotherapy
- 3 Nivo-Ipi (closed to enrollment) (Experimental): Nivolumab plus Ipilimumab
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- 4 Nivo-Ipi-CCNU-TMZ (Experimental): Nivolumab plus Ipilimumab plus Lomustine (CCNU) plus 5-day Temozolomide
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: 5-day Temozolomide; Drug: Lomustine
- 5 Nivo-Ipi-TMZ (Experimental): Nivolumab plus Ipilimumab plus 5-day Temozolomide
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: 5-day Temozolomide
- 6 Nivo-Ipi-Bev-TMZ (Experimental): Nivolumab plus Ipilimumab plus Bevacizumab plus 5-day Temozolomide
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Bevacizumab; Drug: 5-day Temozolomide

INTERVENTIONS:
Drug: Temozolomide — concomitant and 5-day adjuvant temozolomide
  Other Names: temodar
  Arms: 1 SOC (closed to enrollment)
Radiation: conformal brain radiation therapy — standard radiation therapy for newly diagnosed glioblastoma
  Arms: 1 SOC (closed to enrollment)
Drug: Nivolumab — nivolumab 240 mg IV every 2 weeks for the first 28-day cycle, then option to modify to 480 mg IV every 4 weeks
  Other Names: opdivo
  Arms: 3 Nivo-Ipi (closed to enrollment); 4 Nivo-Ipi-CCNU-TMZ; 5 Nivo-Ipi-TMZ; 6 Nivo-Ipi-Bev-TMZ
Drug: Ipilimumab — ipilimumab 1 mg/kg IV every 6 weeks (or every 8 weeks when nivolumab is administered every 4 weeks) for a maximum of 4 doses
  Other Names: yervoy
  Arms: 3 Nivo-Ipi (closed to enrollment); 4 Nivo-Ipi-CCNU-TMZ; 5 Nivo-Ipi-TMZ; 6 Nivo-Ipi-Bev-TMZ
Drug: Bevacizumab — bevacizumab 5 mg/kg IV every 2 weeks (up to 10 mg/kg at treating physician's discretion)
  Other Names: avastin
  Arms: 6 Nivo-Ipi-Bev-TMZ
Drug: 5-day Temozolomide — 150 mg/m^2 oral, once daily on Days 1-5 of each 28-day cycle (stepwise titration every cycle up to 200 mg/m^2 permitted)
  Other Names: temodar
  Arms: 5 Nivo-Ipi-TMZ; 6 Nivo-Ipi-Bev-TMZ
Drug: 5-day Temozolomide — 100 mg/m^2 oral, once daily on Days 2-6 of each 6 week course (stepwise titration every cycle up to 200 mg/m^2 permitted)
  Other Names: temodar
  Arms: 4 Nivo-Ipi-CCNU-TMZ
Drug: Lomustine — 100 mg/m^2 oral, on Day 1 of each 6 week course
  Other Names: CCNU
  Arms: 4 Nivo-Ipi-CCNU-TMZ
Drug: Nivolumab monotherapy — nivolumab 300 mg IV every 2 weeks for the first 28-day cycle, then option to modify to 480 mg IV every 4 weeks
  Other Names: opdivo
  Arms: 2 Nivo

SUMMARY:
The purpose of this study is to test the safety and tolerability of the research study drugs nivolumab, ipilimumab, lomustine, bevacizumab, and temozolomide when used following surgery and before standard therapy with radiation and temozolomide in patients with newly diagnosed high grade glioma.

Additional aims of the study are to:

* Find out side effects (good and bad) of study drug combinations.
* Evaluate any preliminary evidence of anticancer activity of study drug combinations .
* Evaluate tumor characteristics by collecting brain tumor tissue samples.
* Measure the amount of nivolumab and ipilimumab in biospecimens.
* Look at biomarkers in biospecimens.

DETAILED DESCRIPTION:
Patients having a clinically planned surgical procedure (biopsy or cytoreduction) for a suspected diagnosis of high grade glioma will be approached for participation in this study. Tumor tissue obtained from surgery will be used for histological diagnosis and clinical molecular profiling, and excess tumor tissue will be collected for potential correlative studies. A small sample of blood and CSF for research will also be collected.

Once a diagnosis of high grade glioma is confirmed, the patient will be allocated to one of the study arms. Treatment will be started approximately 7-42 days following surgery once the patient has recovered from surgery. Routine clinical evaluations will be performed prior to treatment initiation and throughout treatment as clinically indicated. Radiographic brain imaging will be performed approximately 21-42 after treatment initiation and then routinely for medical management. Tumor response will be assessed according to immunotherapy Response Assessment in Neuro-Oncology (iRANO) Working Group criteria.

Treatment may continue until the patient experiences unacceptable toxicity or clear disease progression. The determination of whether to stop treatment due to disease progression will be based on the investigator's evaluation of the patient's clinical and radiographic condition, taking into consideration the interpretation of localized inflammatory responses that can mimic radiographic features of tumor progress. Patients discontinuing treatment will have further medical management as directed by their treating physician.

As part of follow-up, if the patient undergoes a surgery, results of clinical molecular profiling will be collected, and excess resected tumor tissue will be collected if available along with blood and CSF for correlative studies. A record of any additional anti-cancer treatments and survival status will be made every three to six months.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has the ability to understand and the willingness to provide a signed and dated informed consent form.
2. Participant has the willingness to comply with all study procedures and availability for the duration of the study.
3. Participant is being evaluated for a potential, or known, diagnosis of high grade glioma.
4. Participant is a candidate for brain surgery or has undergone prior surgery and has not received any additional treatment for high grade glioma.
5. Participant is male or female, ≥ 18 years of age.
6. Participant has a Karnofsky Performance Status (KPS) ≥ 60%:

Exclusion Criteria:

1. Participant has received prior anti-cancer treatment for high grade glioma.
2. Participant has a diagnosis of immunodeficiency or active autoimmune disease.
3. Participant is receiving chronic systemic steroid therapy in dosing exceeding 8 mg daily of dexamethasone equivalent or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. Note: This is assessed after surgery, prior to starting drug treatment.
4. Participant has received a live vaccine within 28 days prior to the first dose of study agent. Examples of live vaccines include, but are not limited to measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), typhoid vaccine, and intranasal influenza vaccines (e.g., FluMist®).
5. Participant has a severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to receive study intervention (i.e., uncontrolled diabetes, chronic renal disease, chronic pulmonary disease or active, uncontrolled infection, psychiatric illness/social situations that would limit compliance with study requirements).
6. Participant is a female of childbearing potential who is pregnant or nursing.
7. Participant has a history of thrombotic or hemorrhagic stroke or myocardial infarction within 6 months.
8. Participant has a history of intestinal perforations, fistula, hemorrhages, and/or hemoptysis ≤ 6 months prior to first study treatment.
9. Participant has active gastrointestinal bleeding.
10. Participant has uncontrolled hypertension (systolic blood pressure ≥ 160 mm Hg and/or diastolic blood pressure ≥ 90 mm Hg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities | first 28 days of treatment
  treatment-related adverse events that impact administration of treatment

SECONDARY OUTCOMES:
Treatment-related adverse events | approximately 7 months
  Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.03.
Tumor response rates | up to 5 years
  Evidence of anti-tumor activity as measured according to immunotherapy Response Assessment in Neuro-Oncology (iRANO) criteria.
Progression free survival (PFS) | up to 5 years
  The duration of time from start of treatment until objective tumor response.
Overall survival (OS) | up to 5 years
  The duration of time from start of treatment to death.
Levels of immunotherapeutic agents in specimens | approximately 4 months
  Immunotherapeutic drug levels in specimens.
Change in clinical molecular profile of tumor tissue after treatment | approximately 6 months to 1 year
  Comparison of tumor tissue molecular profile generated from before and after study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD, PhD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- Saint John's Cancer Institute, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Complete de-identified patient data set will be available upon reasonable request to the principal investigator.
Time Frame: beginning one year after completion of the trial (no end date)
Access Criteria: Reasonable request

REFERENCES:
- [Derived] Kesari S, Wojcinski A, Pabla S, Seager RJ, Gill JM, Carrillo JA, Wagle N, Park DJ, Nguyen M, Truong J, Takasumi Y, Chaiken L, Chang SC, Barkhoudarian G, Kelly DF, Juarez TM. Pre-radiation Nivolumab plus ipilimumab in patients with newly diagnosed high-grade gliomas. Oncoimmunology. 2024 Dec 31;13(1):2432728. doi: 10.1080/2162402X.2024.2432728. Epub 2024 Nov 21. PMID 39572979